CLINICAL TRIAL: NCT00878943
Title: A Local, Multi-centre, Open Label Access Study, To Provide Sildenafil Therapy To Eligible Adult Patients With Pulmonary Arterial Hypertension Completing A1481244 Study In India Or Ongoing In A1481269 Study Who Continue To Receive Benefit From Sildenafil Therapy.
Brief Title: Open Label Access Study Of Sildenafil In Adult Patients With Pulmonary Arterial Hypertension Completing A1481244 Study
Acronym: UK 92480
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481269
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Open label access; sildenafil; pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil citrate — 20 mg tablet to be taken thrice daily for 1 year

SUMMARY:
In an earlier study, sildenafil citrate administered to patients of PAH led to improvement in pulmonary arterial pressure, cardiac output, quality of life, and other parameters as compared to placebo. This protocol provides mechanism for patients who have clinical deterioration on other PAH approved therapies to have access to sildenafil prior to marketing authorization in India.

ELIGIBILITY:
Inclusion Criteria:

* Subject who complete the A1481244 study and require Sildenafil (Revatio TM) 20 mg TID therapy.
* All women of childbearing potential must use adequate contraception throughout the study and four weeks after completion of the study

Exclusion Criteria:

* Pregnant or lactating women
* Participation in other studies during study participation
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- India (5):
  - The Institute of Medical Sciences, CARE Hospital, Hyderabad, Andhra Pradesh
  - Mehta Hospital & Cardiopulmonary Care Center, Ahmedabad, Gujarat
  - Bankers Heart Institute, Vadodara, Gujarat
  - St Johns Medical College Hospital, Bangalore, Karnataka
  - Metro Multispeciality Hospital, Noida, Uttar Pradesh

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481269&StudyName=Open%20Label%20Access%20Study%20Of%20Sildenafil%20In%20Adult%20Patients%20With%20Pulmonary%20Arterial%20Hypertension%20Completing%20A1481244%20Study